CLINICAL TRIAL: NCT06070909
Title: Selective Activation of the Infraspinatus During External Rotation Exercises in Participants With Rounded Shoulder Posture: Comparison of 3 Common Exercises and Muscle Architecture-Based Exercise
Brief Title: Selective Activation of the Infraspinatus During External Rotation Exercises in Participants With Rounded Shoulder Posture
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 38b5558f4bdd45f8
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Disease
Keywords: Infraspinatus; Muscle architecture; Rounded Shoulder Posture; Superficial EMG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: The EMG activations — The EMG activations of the middle trapezius, posterior deltoid and infraspinatus muscles in the dominant limb were recorded during exercises in standing external rotation (SER), side-lying position (SDER), scapular plane (SPER) and muscle architecture-based (MABER) positions

SUMMARY:
The purpose of this prospective, cross-sectional study was to evaluate the selective activation of the infraspinatus during external rotation exercises in participants with rounded shoulder postures and compare the different exercise positions. The fifteen (7 males and 8 females) participants with rounded shoulder posture were recruited for this study. The EMG activations of the middle trapezius, posterior deltoid and infraspinatus muscles in the dominant limb were recorded during exercises in standing external rotation (SER), side-lying position (SDER), scapular plane (SPER) and muscle architecture-based (MABER) positions.

ELIGIBILITY:
Inclusion Criteria:

* without shoulder pain,
* totally able to perform overhead activities with no pain or discomfort,
* without a history of shoulder injuries
* with rounded shoulder posture

Exclusion Criteria:

* a history of shoulder muscle injury
* bone fractures in shoulder region
* luxation or subluxation
* cervical dysfunction radiating to upper limbs
* neurologic or musculoskeletal disorders that would prevent shoulder external rotation in the testing postures.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fifteen (7 males and 8 females) participants without shoulder pain, totally able to perform overhead activities with no pain or discomfort, without a history of shoulder injuries, and with rounded shoulder posture were recruited for this study.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
The EMG activations of the middle trapezius, posterior deltoid and infraspinatus muscles in the dominant limb | 4 weeks
  The EMG activations of the middle trapezius, posterior deltoid and infraspinatus muscles in the dominant limb were recorded during exercises in standing external rotation (SER), side-lying position (SDER), scapular plane (SPER) and muscle architecture-based (MABER) positions

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided